CLINICAL TRIAL: NCT00486356
Title: A Phase I Trial of Epirubicin, Carboplatin and Capecitabine in Adult Cancer Patients
Brief Title: Capecitabine, Epirubicin, and Carboplatin in Treating Patients With Progressive, Unresectable, or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0284-04-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Liver Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent gastric cancer; stage IV gastric cancer; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent gallbladder cancer; unresectable gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Capecitabine; Carboplatin; Epirubicin; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- Capecitabine, Epirubicin, and Carboplatin (Experimental): Determine the recommended phase II dose of capecitabine when given together with epirubicin and carboplatin in treating patients with progressive, unresectable, or metastatic cancer.
  Interventions: Drug: capecitabine; Drug: carboplatin; Drug: epirubicin hydrochloride; Genetic: microarray analysis; Genetic: polymorphism analysis; Other: pharmacological study

INTERVENTIONS:
Drug: capecitabine
  Other Names: Xeloda
Drug: carboplatin
  Other Names: Paraplatin
Drug: epirubicin hydrochloride
  Other Names: Ellence
Genetic: microarray analysis
Genetic: polymorphism analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, epirubicin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of capecitabine when given together with epirubicin and carboplatin in treating patients with progressive, unresectable, or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended phase II dose of capecitabine when given together with epirubicin hydrochloride and carboplatin in patients with progressive, unresectable, or metastatic cancer.
* Determine the toxicities of this regimen in these patients.

Secondary

* Correlate end-of-infusion levels of epirubicin hydrochloride and its metabolites with epirubicin hydrochloride dose and clinical toxicity in these patients.
* Correlate the pharmacokinetics of capecitabine with clinical toxicity in these patients.
* Determine the possible correlation between polymorphisms in the promoter region of the thymidylate synthase gene with clinical toxicity in these patients.
* Document antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of capecitabine.

Patients receive epirubicin hydrochloride IV over 2 hours and carboplatin IV over 30 minutes on day 1 and oral capecitabine twice daily on days 2-5, 8-12, and 15-19. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Peripheral blood is collected for pharmacokinetic and pharmacogenetic studies before beginning study treatment and periodically during study. Samples for the pharmacogenetic studies are analyzed for correlation between polymorphisms in the promoter region of the thymidylate synthase gene and clinical toxicity. Patients also undergo bone marrow aspirate before beginning study treatment for molecular profiling studies.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed cancer, meeting 1 of the following criteria:

  * Disease that has progressed on standard therapy
  * Locally advanced but unresectable primary or recurrent solid tumor
  * Metastatic disease, including previously untreated metastatic disease for which study regimen represents reasonable initial chemotherapy with palliative intent (e.g., metastatic gastric cancer, hepatobiliary cancer, or cancer for which no effective standard therapy exists)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* alanine aminotransferase (ALT) & aspartate aminotransferase (AST) ≤ 2.5 times ULN
* Creatinine ≤ 1.6 mg/dL
* Left ventricular ejection fraction ≥ 50%
* Fertile patients must use effective contraception
* Recovered from prior therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) or immunotherapy
* At least 2 weeks since prior radiotherapy
* At least 8 weeks since prior strontium therapy
* At least 4 weeks since prior and no concurrent sorivudine or brivudine

Exclusion Criteria:

* No other potentially curative treatment options available (e.g., surgery, radiotherapy, chemoradiotherapy, or combination chemotherapy)
* No leukemia or lymphoma
* No primary central nervous system (CNS) malignancies or CNS metastases
* No other medical illness that would preclude study treatment
* No active infection requiring IV antibiotic therapy unless the infection has resolved
* No history of allergy to platinum compounds, mannitol, or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* No history of unexpectedly severe intolerance to fluorouracil
* Not pregnant or nursing/negative pregnancy test
* No prior doxorubicin at cumulative doses > 300 mg/m²
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent cimetidine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-01-01 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of capecitabine | Every 28-days until first documented progression up to 63 months
  Establish a recommended Phase II dose of oral capecitabine given twice daily on days 2-5, 8-12, and 15-19 in combination with fixed IV doses of epirubicin and carboplatin given day 1 of each 28-day cycle
Toxicities of combined chemotherapy regimen | Every 28-days until first documented progression up to 63 months
  Evaluate all toxicities associated with this combination chemotherapy regimen: 1 - mild, 2 - moderate, 3 = severe and 4 - life-threatening

SECONDARY OUTCOMES:
End-of-infusion levels of epirubicin hydrochloride/metabolites and incidence of correlation with epirubicin hydrochloride dosing and clinical toxicity | Each day of dosing up to 63 months
  Correlation of end-of-infusion levels of epirubicin hydrochloride and its metabolites with epirubicin hydrochloride dosing and clinical toxicity (1 - mild, 2 - moderate, 3 = severe and 4 - life-threatening)
Correlation of the pharmacokinetics (speed of appearance in the blood plasma and its concentration) of capecitabine with clinical toxicity | Each day of dosing up to 63 months
  Measure the pharmacokinetics of capecitabine and correlate these parameters with clinical toxicity
Incidence of Correlation between polymorphisms in the promoter region of the thymidylate synthase gene with clinical toxicity | Post-treatment up to 63 months
  Assess possible correlation between polymorphisms in the promoter region of the thymidylate synthase gene with clinical toxicity
Antitumor activity | Prior to cycle 1, and then every two 28 day cycles up to 63 months
  Document any anti-tumor activity (MTT assay is a quantitative and sensitive detection of cell proliferation as it measures the growth rate of cells by virtue of a linear relationship between cell activity and absorbance.)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Grem, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Eppley Cancer Center, Omaha, Nebraska, United States